CLINICAL TRIAL: NCT02869438
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase 3b Study to Evaluate the Onset of Effect and Time Course of Change in Lung Function With Benralizumab in Severe, Uncontrolled Asthma Patients With Eosinophilic Inflammation
Brief Title: A Study to Evaluate the Onset of Effect and Time Course of Change in Lung Function With Benralizumab in Severe, Uncontrolled Asthma Patients With Eosinophilic Inflammation
Acronym: SOLANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D3250C00038; 2016-002094-36 (EudraCT Number); U1111-1185-6625 (Other: WHO (UTN number))
Record Dates: First submitted 2016-08-16; First posted 2016-08-17 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benralizumab arm (Experimental): Benralizumab administered subcutaneously
  Interventions: Drug: Benralizumab
- Placebo arm (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Benralizumab — Benralizumab administered subcutaneously at Visit 1 (Day 0), Visit 8 (Day28 +/- 3 days) and Visit 9 (Day 56 +/- 3 days)
  Arms: Benralizumab arm
Other: Placebo — Placebo administered subcutaneously at Visit 1 (Day 0), Visit 8 (Day28 +/- 3 days) and Visit 9 (Day 56 +/- 3 days)
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to investigate the onset and maintenance of effect of benralizumab on lung function, blood eosinophils, asthma control metrics and quality of life during 12-week treatment in patients with uncontrolled, severe asthma with eosinophilic inflammation. A subset of patients will take part in body plethysmography substudy to further investigate the effect on lung function.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent for study participation must be obtained prior to any study related procedures being performed and according to international guidelines and/or applicable European Union (EU) guidelines.
2. Female and male aged 18 to 75 years inclusively at the time of Visit 1
3. Documented current treatment with ICS and LABA for at least 30 days prior to Visit 1. The ICS and LABA can be parts of a combination product or given by separate inhalers. The ICS dose must be greater than or equal to 500 μg/day fluticasone propionate dry powder formulation or equivalent daily. Additional asthma controller medications, eg, oral corticosteroids, long-acting antimuscarinics (LAMAs), LTRAs, theophylline etc. are allowed if they have been used for at least 30 days prior to Visit 1
4. History of at least 2 asthma exacerbations that required treatment with systemic corticosteroids (intramuscular (IM), intravenous (IV), or oral) in the 12 months prior to Visit 1. For patients receiving corticosteroids as a maintenance therapy, the corticosteroid treatment for the exacerbation is defined as a temporary increase of their maintenance dose.
5. Pre-bronchodilator (pre-BD) FEV1 of < 80% predicted at Visit 2 or Visit 3
6. ACQ-6 score ≥1.5 at Visit 1
7. Evidence of asthma as documented by airway reversibility (FEV1 ≥12% and 200 ml) demonstrated at Visit 1, Visit 2 or Visit 3. For patients entering the body plethysmography sub-study, reversibility must be demonstrated at Visit 1 or at Visit 2 only
8. Peripheral blood eosinophil count of ≥300 cells/μL assessed by central lab at Visit 1
9. Women of childbearing potential (WOCBP) must use an effective form of birth control confirmed by the Investigator. WOCBP must also have negative serum pregnancy test result on Visit 1.

   Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomization without an alternative medical cause. The following agespecific requirements apply:
   * Women <50 years old are considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
   * Women ≥50 years old are considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
10. All male patients who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of IP until 16 weeks after their last dose
11. Weight of ≥40 kg

Additional inclusion criteria applicable for the Body Plethysmography substudy 1.Residual volume ≥125% of predicted at Visit 3.

Inclusion criteria at randomization visit

1. At least 1 of the following within 7 days prior to randomization:

   * Daytime or nighttime asthma symptoms for 2 or more days;
   * Rescue SABA use for 2 or more days;
   * Nighttime awakenings due to asthma at least 1 night during the 7-day period
2. ACQ >0.75 at Visit 4 prior to randomization.
3. A negative urine pregnancy test in WOCBP prior to administration of IP

Exclusion criteria

1. Clinically important pulmonary disease other than asthma (eg, active lung infection, COPD, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome)
2. Life-threatening asthma defined as episodes requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episodes within the 12 months prior to Visit 1.
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period
4. An upper respiratory tract infection or an asthma exacerbation that required treatment with systemic corticosteroids or an increase in regular maintenance dose of OCS during the screening/run-in period prior to randomization Visit 4
5. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study
6. Known history of allergy or reaction to any component of the investigational product formulation
7. History of anaphylaxis to any biologic therapy
8. History of Guillain-Barré syndrome
9. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy
10. Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study
11. Any clinically significant cardiac disease or any electrocardiogram (ECG) abnormality obtained during the screening/run-in period, which in the opinion of the Investigator may put the patient at risk or interfere with study assessments
12. History of alcohol or drug abuse within 12 months prior to the date informed consent is obtained
13. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Patients with a history of hepatitis B vaccination without history of hepatitis B are allowed to enroll
14. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test
15. Current smokers or former smokers with a smoking history of ≥10 pack years. A former smoker is defined as a patient who quit smoking at least 6 months prior to Visit 1
16. Current malignancy, or history of malignancy, except for:

    * Patients who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained.
    * Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.
17. Use of immunosuppressive medication (including but not limited to: oral corticosteroids [for reasons other than asthma], methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroids or any experimental anti-inflammatory therapy) within 3 months prior to the date informed consent
18. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥1.5 times the upper limit of normal (ULN) confirmed during screening period
19. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained
20. Receipt of any marketed (eg, omalizumab, mepolizumab etc.) or investigational biologic within 4 months or 5 half-lives prior to the date informed consent is obtained, whichever is longer
21. Receipt of live attenuated vaccines 30 days prior to the date of randomization
22. Receipt of any investigational medication within 30 days or 5 half-lives prior to randomization, whichever is longer
23. Previously received benralizumab (MEDI-563)
24. Planned surgical procedures during the conduct of the study
25. Currently breastfeeding or lactating women
26. Previous randomization in the present study
27. Concurrent enrolment in another interventional or post-authorization safety study (PASS).
28. AstraZeneca staff involved in the planning and/or conduct of the study
29. Employees of the study center or any other individuals involved with the conduct of the study or immediate family members of such individuals

Exclusion criteria at randomization Visit 4

1. Greater than/equal to 20% change in mean Pre BD FEV1 value at randomization Visit 4 from the mean pre BD FEV1 calculated from the pre BD FEV1 recorded at Visit 2 and Visit 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reynold A Panettieri, Doctor of Medicine, Principal Investigator — Child Health Institute of NJ, 89 French Street, Suite 4210, New Brunswick, NJ, 08901, USA
Locations (42):
- United States (16):
  - Research Site, Scottsboro, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Denver, Colorado
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Rochester, Minnesota
  - Research Site, New Bern, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Lampasas, Texas
  - Research Site, McKinney, Texas
- Chile (2):
  - Research Site, Curicó
  - Research Site, Santiago
- Germany (8):
  - Research Site, Bamberg
  - Research Site, Darmstadt
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, München
- Hungary (8):
  - Research Site, Balassagyarmat
  - Research Site, Edelény
  - Research Site, Farkasgyepü
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Komárom
  - Research Site, Miskolc
  - Research Site, Pécs
- Philippines (4):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Manila
  - Research Site, Quezon City
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seoul

REFERENCES:
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4080&filename=d3250c00038-csp-v1_Redacted.pdf
- See also: SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4080&filename=d3250c00038-sap-ed-2_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 233 participants were randomized to receive treatment in study D3250C00038 (Solana) with benralizumab 30 mg or placebo. Of the 233 patients randomised, all (100.0%) received treatment with study drug. 118 (50.6%) patients received benralizumab 30 mg and 115 (49.4%) patients received placebo.
Groups:
- Benra 30 mg: 12-week treatment period and receive Benra 30 mg at Day 0, Day 28 (±3 days), and Day 56 (±3 days).
- Placebo: 12-week treatment period and receive Placebo at Day 0, Day 28 (±3 days), and Day 56 (±3 days).
Period: Overall Study
Arm/Group | Benra 30 mg | Placebo
Started | 118 | 115
Completed | 115 | 113
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benra 30 mg | Placebo | Total
Number analyzed (Participants) | 118 | 115 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (13.62) | 50.9 (12.34) | 51.4 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 83 | 157
  Male | 44 | 32 | 76
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 69 | 67 | 136
  Black or African American | 3 | 4 | 7
  Asian | 39 | 40 | 79
  Other | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 4) to Day 28 (Visit 8), Day 56 (Visit 9), and Day 84 (Visit 10) in Pre-BD FEV1
Description: The average over the mean differences between benralizumab and placebo for change from baseline in pre-BD FEV1 is used to determine if the study is positive and to determine maintenance of effect. The first post baseline time point where the p-value for the mean difference between benralizumab and placebo is less than or equal to 0.05 is used to determine time to onset of effect.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Liter
  Day 28: number analyzed (Participants) | 118 | 113
  Day 28 | 0.21 (0.335) | 0.132 (0.316)
  Day 56: number analyzed (Participants) | 116 | 113
  Day 56 | 0.22 (0.367) | 0.203 (0.349)
  Day 84: number analyzed (Participants) | 114 | 114
  Day 84 | 0.209 (0.344) | 0.149 (0.366)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0707, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [-0.007 to 0.161] — For Day 28
Statistical Analysis 2: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.7747, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.077 to 0.104] — For Day 56
Statistical Analysis 3: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0969, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.014 to 0.173] — For Day 84
Statistical Analysis 4: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.1558, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [-0.022 to 0.135] — For average over Day 28, 56, and 84

2. Primary Outcome: Change From Baseline (Visit 4) to End of Treatment Day 84 (Visit 10) in Residual Volume (RV)
Description: Body plethysmography was performed for sub-study patients. Lung volume subdivisions measures were performed by the investigator or qualified designee according to ATS/ERS guidelines.
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
Liter | -0.415 (0.609) | -0.208 (0.528)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.2847, Mixed Models Analysis; Model includes covariates of treatment, baseline RV, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.176, 95% CI 2-sided [-0.505 to 0.153]

3. Secondary Outcome: Percent Change From Baseline to End of Treatment in Eosinophils Counts
Description: Percent change from baseline to Day 84
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Percent change | -88.55 [-100 to -12.5] | 11.55 [-91.4 to 833.3]
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Model includes covariates of treatment, baseline eosinophils counts, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -101.0, 95% CI 2-sided [-118.9 to -83.06]

4. Secondary Outcome: Change From Baseline (Visit 4) to Post Baseline Visits in Pre-BD FEV1
Description: Post baseline visits include Day 3, Day 7, Day 14, Day 28, Day 56, Day 84. [Note: Day 28, 56, 84 are presented in the Primary measure.]
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Liter
  Day 3: number analyzed (Participants) | 110 | 107
  Day 3 | 0.104 (0.223) | 0.081 (0.269)
  Day 7: number analyzed (Participants) | 118 | 112
  Day 7 | 0.125 (0.229) | 0.081 (0.263)
  Day 14: number analyzed (Participants) | 118 | 113
  Day 14 | 0.126 (0.3) | 0.1 (0.287)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.6384, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.015, 95% CI 2-sided [-0.049 to 0.08] — For Day 3
Statistical Analysis 2: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.148, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [-0.016 to 0.109] — For Day 7
Statistical Analysis 3: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.4959, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.049 to 0.101] — For Day 14

5. Secondary Outcome: Change From Baseline to Post Baseline for Pre-BD FVC
Description: Post baseline visits include Day 3, Day 7, Day 14, Day 28, Day 56, and Day 84.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Liter
  Day 3: number analyzed (Participants) | 110 | 107
  Day 3 | 0.122 (0.247) | 0.11 (0.267)
  Day 7: number analyzed (Participants) | 118 | 112
  Day 7 | 0.138 (0.277) | 0.099 (0.292)
  Day 14: number analyzed (Participants) | 118 | 113
  Day 14 | 0.126 (0.331) | 0.111 (0.312)
  Day 28: number analyzed (Participants) | 118 | 113
  Day 28 | 0.21 (0.347) | 0.134 (0.34)
  Day 56: number analyzed (Participants) | 116 | 113
  Day 56 | 0.211 (0.404) | 0.187 (0.369)
  Day 84: number analyzed (Participants) | 114 | 114
  Day 84 | 0.213 (0.376) | 0.131 (0.359)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.8667, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.062 to 0.073] — For Day 3
Statistical Analysis 2: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.2734, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.041, 95% CI 2-sided [-0.033 to 0.115] — For Day 7
Statistical Analysis 3: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.7252, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.015, 95% CI 2-sided [-0.068 to 0.098] — For Day 14
Statistical Analysis 4: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0976, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [-0.014 to 0.164] — For Day 28
Statistical Analysis 5: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.6536, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.077 to 0.122] — For Day 56
Statistical Analysis 6: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0595, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.092, 95% CI 2-sided [-0.004 to 0.188] — For Day 84
Statistical Analysis 7: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.1377, Mixed Models Analysis; Model includes covariates of treatment, baseline pre-BD FVC, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [-0.02 to 0.147] — For average of Day 28, 56, 84

6. Secondary Outcome: Percentage of Pre-BD FEV1 Responder
Description: Pre-BD FEV1 responder is defined as change from baseline in FEV1 >=100 ml
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Percentage of Participants
  Day 3: number analyzed (Participants) | 110 | 107
  Day 3 | 48.2 | 37.4
  Day 7: number analyzed (Participants) | 118 | 112
  Day 7 | 48.3 | 42.0
  Day 14: number analyzed (Participants) | 118 | 113
  Day 14 | 50.0 | 38.9
  Day 28: number analyzed (Participants) | 118 | 113
  Day 28 | 57.6 | 46.9
  Day 56: number analyzed (Participants) | 116 | 113
  Day 56 | 62.1 | 55.8
  Day 84: number analyzed (Participants) | 114 | 114
  Day 84 | 57.9 | 51.8
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.1604, Regression, Logistic; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.85 to 2.58] — For Day 3
Statistical Analysis 2: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.3400, Regression, Logistic; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.76 to 2.19] — For Day 7
Statistical Analysis 3: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0924, Regression, Logistic; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.93 to 2.70] — For Day 14
Statistical Analysis 4: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.1052, Regression, Logistic; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.91 to 2.71] — For Day 28
Statistical Analysis 5: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.3271, Regression, Logistic; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.77 to 2.21] — For Day 56
Statistical Analysis 6: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.3017, Regression, Logistic; Model includes covariates of treatment, baseline pre-BD FEV1, region, visit, treatment by visit interaction; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.77 to 2.29] — For Day 84

7. Secondary Outcome: Change From Baseline in ACQ-6
Description: ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses. Mean scores of <=0.75 indicates well-controlled asthma, scores between 0.75 to <=1.5 indicate partly controlled asthma, and >1.5 indicates not well controlled asthma.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Score on a scale
  Day 14: number analyzed (Participants) | 118 | 113
  Day 14 | -0.989 (0.901) | -0.665 (0.837)
  Day 28: number analyzed (Participants) | 118 | 113
  Day 28 | -1.126 (0.947) | -0.693 (0.869)
  Day 56: number analyzed (Participants) | 115 | 113
  Day 56 | -1.164 (1.132) | -0.827 (1.023)
  Day 84: number analyzed (Participants) | 114 | 113
  Day 84 | -1.355 (1.146) | -0.867 (1.114)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0024, Mixed Models Analysis; Model includes covariates of treatment, baseline ACQ-6 score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.293, 95% CI 2-sided [-0.481 to -0.105] — For Day 14
Statistical Analysis 2: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Model includes covariates of treatment, baseline ACQ-6 score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.402, 95% CI 2-sided [-0.609 to -0.195] — For Day 28
Statistical Analysis 3: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0117, Mixed Models Analysis; Model includes covariates of treatment, baseline ACQ-6 score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.312, 95% CI 2-sided [-0.554 to -0.07] — For Day 56
Statistical Analysis 4: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Model includes covariates of treatment, baseline ACQ-6 score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.472, 95% CI 2-sided [-0.731 to -0.213] — For Day 84
Statistical Analysis 5: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Model includes covariates of treatment, baseline ACQ-6 score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.395, 95% CI 2-sided [-0.603 to -0.188] — For average of Day 28, 56, 84

8. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is designed to measure health impairment in patients with asthma and COPD. It contains two parts: Part 1 (Questions 1 to 8) covers the patients' recollection of their symptoms over a preceding 4 weeks; Part 2, 42 items, relates to the daily activity and psychosocial impacts of the individual's respiratory condition. Total score is presented as a percentage of overall impairment, in which 100 represents the worst possible health status, while 0 indicates the best.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Score on a scale
  Day 28: number analyzed (Participants) | 118 | 113
  Day 28 | -16.956 (15.51) | -9.444 (14.136)
  Day 56: number analyzed (Participants) | 115 | 113
  Day 56 | -19.941 (21.528) | -13.802 (16.705)
  Day 84: number analyzed (Participants) | 114 | 113
  Day 84 | -23.343 (20.302) | -14.385 (18.836)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Model includes covariates of treatment, baseline SGRQ score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -7.229, 95% CI 2-sided [-10.832 to -3.626] — For Day 28
Statistical Analysis 2: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0115, Mixed Models Analysis; Model includes covariates of treatment, baseline SGRQ score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -5.942, 95% CI 2-sided [-10.538 to -1.346] — For Day 56
Statistical Analysis 3: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Model includes covariates of treatment, baseline SGRQ score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -8.599, 95% CI 2-sided [-13.3 to -3.898] — For Day 84
Statistical Analysis 4: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Model includes covariates of treatment, baseline SGRQ score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -7.257, 95% CI 2-sided [-11.133 to -3.38] — For average of Day 28, 56, 84

9. Secondary Outcome: Change From Baseline to End of Treatment in FeNO
Description: Airway inflammation was evaluated via fractional exhaled nitric oxide (FeNO) measurement.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
ppb | 5.92 (45.295) | 0.05 (27.634)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.2825, Mixed Models Analysis; Model includes covariates of treatment, baseline FeNO value, region, visit, treatment by visit interaction; Mean Difference (Final Values) = 5.414, 95% CI 2-sided [-4.492 to 15.321]

10. Secondary Outcome: Change From Baseline to End of Treatment in Total Lung Capacity (TLC) for Sub-study Patients
Description: Lung volume subdivisions include total lung capacity (TLC), residual volume (RV), vital capacity (VC), functional residual capacity (FRC), and inspiratory capacity (IC), as well as airway resistance (Raw and SGaw) measurements.
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
Liter | -0.276 (0.677) | -0.175 (0.418)

11. Secondary Outcome: Change From Baseline to End of Treatment in Ratio of Residual Volume (RV) and Total Lung Capacity (TLC) for Sub-study Patients
Description: as for outcome 10
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
ratio | -0.05 (0.056) | -0.026 (0.087)

12. Secondary Outcome: Change From Baseline to End of Treatment in Inspiratory Capacity (IC) for Sub-study Patients
Description: as for outcome 10
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
Liter | 0.119 (0.447) | -0.268 (0.603)

13. Secondary Outcome: Change From Baseline to End of Treatment in Functional Residual Capacity (FRC) for Sub-study Patients
Description: as for outcome 10
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
Liter | -0.394 (0.783) | 0.093 (0.466)

14. Secondary Outcome: Change From Baseline to End of Treatment in Vital Capacity (VC) for Sub-study Patients
Description: as for outcome 10
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
Liter | 0.139 (0.245) | 0.033 (0.676)

15. Secondary Outcome: Duration of IP Administration
Description: Duration of IP administration is last IP dose date - first IP dose +1.
Time Frame: From first IP to last IP
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Days | 55.9 (7.83) | 56.2 (7.61)

16. Other Pre Specified Outcome: Serum Concentration of Benralizumab
Description: PK sample was collected pre-dose at each visit
Time Frame: From first dose to end of treatment period (Day 84)
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 117
ng/mL
  Baseline: number analyzed (Participants) | 116
  Baseline | 1.95 (NA) — Only 1 patient had PK concentration detectable, ie, PK concentration <LLOQ for 115 participants.
  Day 3: number analyzed (Participants) | 91
  Day 3 | 1266.78 (199.59)
  Day 7: number analyzed (Participants) | 112
  Day 7 | 1449.47 (125.02)
  Day 14: number analyzed (Participants) | 116
  Day 14 | 1317.92 (79.53)
  Day 28: number analyzed (Participants) | 114
  Day 28 | 738.47 (80.77)
  Day 56: number analyzed (Participants) | 114
  Day 56 | 1015.72 (59.74)
  Day 84: number analyzed (Participants) | 108
  Day 84 | 1079.22 (73.24)

17. Other Pre Specified Outcome: PK Parameter of Benralizumab (Cmax)
Description: PK parameters are derived in patients with at least three qualifiable serum PK concentrations post first dose (collected on Day 3, 7, and either 14, or 28)
Time Frame: First IP dose cycle (ie, data collected on Days 3, 7, 14 and 28)
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 117
ng/mL | 1729.6 (36.8)

18. Other Pre Specified Outcome: Anti-drug Antibody Responses
Description: Anti-drug antibody responses at baseline and post baseline, including nAb responses
Time Frame: From first IP dose to end of treatment period (Day 84)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Participants
  ADA prevalence: number analyzed (Participants) | 117 | 114
  ADA prevalence | 7 | 2
  nAb prevalence: number analyzed (Participants) | 117 | 114
  nAb prevalence | 2 | 0
  Both baseline and post baseline positive: number analyzed (Participants) | 114 | 113
  Both baseline and post baseline positive | 1 | 2
  Only post baseline positive: number analyzed (Participants) | 116 | 113
  Only post baseline positive | 5 | 0
  Only baseline positive: number analyzed (Participants) | 115 | 114
  Only baseline positive | 1 | 0

19. Other Pre Specified Outcome: Change From Baseline to End of Treatment in PGI-S
Description: The patient global impression of severity (PGI-S) is a single item designed to capture the patient's perception of overall symptom severity at the time of the completion using a 6-point categorical response scale (no symptom [0] to very severe symptom [5])
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Score on a scale | -1.2 (1.31) | -0.8 (1.21)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Test type: Superiority; p = 0.0120, Mixed Models Analysis; Model includes covariates of treatment, baseline PGI-S score, region, visit, treatment by visit interaction; Mean Difference (Final Values) = -0.365, 95% CI 2-sided [-0.649 to -0.081] — For Day 84

20. Other Pre Specified Outcome: Change From Baseline to End of Treatment in CGI-C
Description: Clinician global impression of change (CGI-C) is used for an overall evaluation of response to treatment. The investigator is asked to rate the degree of change in overall asthma status compare to the start of treatment. A 7-point rating scale is used from 1=very much improved to 7=very much worse.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Participants
  Very much improved | 18 | 10
  Much improved | 39 | 36
  Minimally improved | 39 | 28
  No change | 17 | 28
  Minimally worse | 0 | 7
  Much worse | 0 | 1
  Very much worse | 0 | 0
  Missing | 5 | 5
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Responder analysis: responder is defined as Very much improved, improved, and minimally improved; Test type: Superiority; p = 0.0018, Regression, Logistic; Model includes covariates of treatment, region; Odds Ratio (OR) = 2.97, 95% CI 2-sided [1.50 to 5.88] — For Day 84

21. Other Pre Specified Outcome: Change From Baseline to End of Treatment in PGI-C
Description: Patient global impression of change (PGI-C) is used for an overall evaluation of response to treatment. The patient is asked to rate the degree of change in overall asthma status compare to the start of treatment. A 7-point rating scale is used from 1=very much improved to 7=very much worse.
Time Frame: From first IP dose to Day 84
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 118 | 115
Participants
  Very much improved | 32 | 17
  Much improved | 42 | 35
  Minimally improved | 23 | 29
  No change | 14 | 27
  Minimally worse | 1 | 4
  Much worse | 1 | 1
  Very much worse | 1 | 0
  Missing | 4 | 2
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; Responder analysis: responder is defined as Very much improved, improved, and minimally improved; Test type: Superiority; p = 0.0107, Regression, Logistic; Model includes covariates of treatment, region; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.24 to 5.09] — For Day 84

22. Other Pre Specified Outcome: Change From Baseline to End of Treatment in Specific Airway Resistance (SGaw) for Sub-study Patients
Description: as for outcome 10
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: 1/(kPa*sec)
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
1/(kPa*sec) | -0.05 (0.146) | 0.052 (0.224)

23. Other Pre Specified Outcome: Change From Baseline to End of Treatment in Airway Resistance (Raw) for Sub-study Patients
Description: as for outcome 10
Time Frame: From first IP dose to Day 84
Population: Body plethysmography sub-study analysis set
Measure: Mean (Standard Deviation); unit: kPa/L/sec
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 18 | 22
kPa/L/sec | -0.233 (1.509) | -0.2 (0.532)

ADVERSE EVENTS:
Time Frame: From informed consent form was signed to end of study (ie, Day 112 follow-up)
Arm/Group | Benra 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/115
Serious Adverse Events (participants affected / at risk) | 1/118 | 7/115
Other Adverse Events (participants affected / at risk) | 28/118 | 30/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=118) | Placebo (N=115)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=118) | Placebo (N=115)
Bronchitis (Infections and infestations) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (9) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 6 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT02869438/SAP_000.pdf
  • Study Protocol (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT02869438/Prot_001.pdf